CLINICAL TRIAL: NCT05306535
Title: Effect of Occlusal Reduction on Relief of Pain and Sensitivity to Percussion in Patients With Irreversible Pulpitis and Symptomatic Apical Periodontitis Treated in a Single Visit- a Randomized Clinical Trial
Brief Title: Effect of Occlusal Reduction on Relief of Pain and Sensitivity to Percussion in Patients With Irreversible Pulpitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Altamash Institute of Dental Medicine (Other)
Responsible Party: Principal Investigator, Hira Abbasi, Principal Investigator, Altamash Institute of Dental Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Endodontic Pain
Record Dates: First submitted 2022-03-15; First posted 2022-04-01 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Post Operative Pain; Post-Op Complication
Keywords: Occlusal reduction
MeSH Terms: conditions — Pain, Postoperative; Postoperative Complications

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- occlusal reduction (Experimental): Performing occlusal reduction on the experimental tooth until absence of occlusal contact is confirmed following completion of the endodontic treatment
  Interventions: Procedure: Occlusal reduction
- control (No Intervention): No occlusal reduction or modification of the occlusal anatomy will be performed

INTERVENTIONS:
Procedure: Occlusal reduction — Occlusal reduction of the experimental single rooted tooth after root canal completion will be done to evaluation reduction in postoperative pain and sensitivity to percussion
  Arms: occlusal reduction

SUMMARY:
One of the most important aspects of endodontic practice is to abate pain during and post root canal treatment. An endodontist by all means should provide a painless endodontic treatment to their patients. This study is carried out to determine the effect of occlusal reduction on relief of pain and percussion in patients with irreversible pulpitis and symptomatic apical periodontitis treated in a single visit root canal treatment. Pain will be assessed preoperatively and then post operatively after completion of the root canal at 6 hours, 12 hours, 24 hours, 48 hours and 72 hours following obturation of root canal.

DETAILED DESCRIPTION:
The objective of this randomized clinical trial is to evaluate the impact of occlusal reduction on the incidence of post obturation pain. 56 patients will be allocated randomly into 2 groups keeping 28 patients in each group which will meet the inclusion criteria of the study, patients diagnosed with symptomatic irreversible pulpitis and symptomatic apical periodontitis and requiring porcelain fused to metal crown with age ranging from 18 to 50 years. In the interventional group 2mm reduction will be done and assessment will be done to confirm the absence of occlusal contact while in control group no modification will be carried out on the occlusal surface. Single visit endodontic treatment will be carried out with 2.5% sodium hypochlorite for disinfection of the canal followed by crown down technique using rotary nickel titanium files for shaping the canals followed by obturating the canals with lateral condensation technique.

Pain will be assessed preoperatively and then post operatively at 6 hours, 12 hours, 24 hours, 48 hours and 72 hours following obturation of root canal. Visual Analogue Scale (VAS) will be used as a primary outcome measure.The VAS consists of a 10-cm line having two extremes NO PAIN and Extreme pain. Patients will be asked to choose the mark that represents their level of pain at the intervals mentioned above . Pain level are assigned to one of four categorical scores

1, None(0); 2, Mild (1-3) ; 3 Moderate (4-6); 4, Severe (7-10) 10. Tenderness to percussion will be evaluated postoperatively at 48 hour with readings either positive to tenderness or negative to tenderness Positive to tenderness will evaluate treatment not effective Negative to tenderness at 48 hour post obturation will evaluate treatment effectiveness Patients will be given placebo for administration in case severe pain and ibuprofen 400mg if the pain persisted. Documentation of intake of either placebo or analgesic will be done by the patient.

ELIGIBILITY:
Inclusion Criteria:

* No medical history
* patients suffering from Symptomatic Irreversible Pulpitis
* patients suffering from Apical Periodontitis
* patients requiring porcelain fused to metal crown

Exclusion Criteria:

* Patients who were not suitable for conventional root canal treatment
* multirooted teeth

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Post Obturation pain | 6 hours upto 48 hours following obturation
  Postobturation pain is measured using the visual analogue scale(VAS) with readings from 0-10 where 0 represents no pain and 10 represents the worst pain measured.
Tenderness to percussion | At 48 hours post completion of the root canal treatment
  Tenderness to percussion will be evaluated (score 0: no pain, score 1: slight pain score 2: severe pain)

SECONDARY OUTCOMES:
Incidence of placebo and analgesic intake | from 6 hours up to 48 hours following completion of root canal
  The incidence of placebo and number analgesic taken will be recorded by the patient

CONTACTS AND LOCATIONS:
Overall Officials: Hira Danish, Principal Investigator — Employee
Locations (1):
- Hira Danish, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No